CLINICAL TRIAL: NCT00996632
Title: Randomized Controlled Study of Benefits of Ultrasonic Knife in Breast Cancer Surgery
Brief Title: The Use of a High-frequency Ultrasonic Knife in Breast Cancer Surgery
Acronym: UKBC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Trieste (Other)
Responsible Party: Pr Nicolò de Manzini, University of Trieste
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MGiuricin
Record Dates: First submitted 2009-04-24; First posted 2009-10-16 (Estimated); Results first posted 2009-10-16 (Estimated); Last update posted 2009-11-11 (Estimated); Status verified 2009-11

CONDITIONS: Breast Cancer
Keywords: breast cancer; ultrasonic knife; volume drainage
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Patients were operated using an ultrasonic knife (Ultracision®, Ethicon Endo Surgery)
  Interventions: Procedure: ultrasonic knife (Ultracision®, Ethicon Endo Surgery)
- B (Active Comparator): Patients were operated using a conventional diarthermy knife
  Interventions: Procedure: conventional diarthermy knife

INTERVENTIONS:
Procedure: ultrasonic knife (Ultracision®, Ethicon Endo Surgery) — mastectomy or quadrantectomy and axillary dissection by an ultrasonic knife (Ultracision®, Ethicon Endo Surgery)
  Arms: A
Procedure: conventional diarthermy knife — mastectomy or quadrantectomy and axillary dissection using conventional diarthermy knife
  Arms: B

SUMMARY:
Background: Lymphatic stasis and seroma formation are common complications of axillary lymphadenectomy in breast cancer surgery. The investigators aim is to test the hypothesis that the use of an ultrasonic knife for axillary dissection reduces the total amount and duration of persistent drainage and length of hospital stay. Method: The investigators have conducted a randomized trial on 94 patients (1 male, 93 females, mean age 64.7 years) who presented to the investigators unit with operable breast carcinoma. Patients in group A (38 cases) were operated on using exclusively the ultrasonic knife. Patients in group B (56 cases) were operated on using the conventional diathermy knife.

DETAILED DESCRIPTION:
The ultrasonic knife we have used in our study exploits the electrical impulses produced by a high-frequency ultrasound generator, transferred to a hand piece and converted into a mechanical movement at a frequency of 55.5 kHz (11,12) (Ultracision®, Ethicon Endo Surgery ). We have chosen this instrument because the relatively low temperatures generated in the process, ranging from 50 to 100 °C, result in a coagulative necrosis which allows both cutting and effective sealing of blood and lymphatic vessels, therefore preventing lymphatic leaks more effectively compared with conventional diathermy. The latter produces temperature up to 400 °C resulting in char formation and deleterious thermal effects to a distance of up to 1cm from the blade and extensive formation of necrotic tissue.

We have estimated Using the data of a previous unpublished pilot study, the sample size required for our trial using the data of a previous unpublished pilot study, indicating that to detect a significant difference in length of stay (delta = 4of four days, with a mean standard deviationsdigma of = 4.5 days, between the two groups with a level of significance of alpha = 5% and a power of1 - beta = 90%), we needed to enroll was estimated in 28 patients in each group arm. As a precaution we decided to increase the sample size by 25% to 35 patients per group arm, in case we needed to use non-parametric tests in subsequent statistical analysis. A total of 94 patients with operable breast carcinoma were recruited between January 2000 and December 2004: 1 male and 93 females (min 34, q1 58, median 65, mean 64.7, q3 73, max 95). All patients underwent total mastectomy or quadrantectomy and 1st or 2nd level axillary lymphadenectomy. Patients were randomly allocated to two treatment groups: patients allocated to Group A were operated on using exclusively the ultrasonic knife (Ultracision®, Ethicon Endo Surgery) for both the mastectomy or quadrantectomy and axillary dissection (38 cases, mean age of 64.6 years, min 34, q1 58, median 66, q3 70, max 95); patients allocated to Group B (control group) were operated on using a conventional diarthermy knife was (56 cases, mean age of 65.0 years,min 37, q1 59, median 65, q3 74, max 89). In all cases the type of a redon n°14 suction drain was left in the axillary cavity and removed as soon as the amount of fluid dropped to 35 ml/24h or less. The patient was discharged home the same day the drain was removed.

During the postoperative period the following data were collected: the total amount of fluid drained, the number of days the drain was leftof drainage, the length of post-operative stay, and early and late complications. Early complications were specifically recorded: wound seromas and hematomas, wound infections, necrosis of wound margins and period of time (in days) the seroma needed to be needle-aspirated following removal of the drain. Late complications recorded were lymphedema, strength and sensation deficits and chronic arm pain. A cost analysis was also done considering materials employed and length of hospital stay. Statistical analysis was done using open source "R" software, version 2.5.1 (18). The Shapiro-Wilk test was used to verify the normal distribution of data; heteroscedastic, normally distributed data were analysed using the F-test of variance; Student's t test was used for homoscedastic data. For non normally distributed data the non-parametric Wilcoxon-Mann-Whitney test was used. Survival analysis was analysed using Cox's regression model, in the hypothesis of proportional risk.

ELIGIBILITY:
Inclusion Criteria:

* Operable breast cancer

Exclusion Criteria:

* Inoperable breast cancer
* BMI > 25
* Neoadiuvant radioterapy
* Carcinomastitis
* Previous phlebitis of omolateral arm
* Collagen disease

Ages: 36 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2000-09; Primary Completion 2004-09 (Actual); Study Completion 2004-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolò de Manzini, Professor, Principal Investigator — University of Trieste
Locations (2):
- Italy (2):
  - University of Trieste, Trieste, Trieste
  - University of Trieste, Trieste

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients affected by Breast Cancer
Groups:
- Ultrasonic: Patients were operated using an ultrasonic knife (Ultracision Ethicon TM)
- Conventional: Patients were operated by a conventional diatherm knife
Period: Overall Study
Arm/Group | Ultrasonic | Conventional
Started | 38 | 56
Completed | 38 | 56
Not Completed | 0 | 0
Not completed — Physician Decision | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ultrasonic | Conventional | Total
Number analyzed (Participants) | 38 | 56 | 94
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 26 | 45
  >=65 years | 19 | 30 | 49
Age Continuous [Mean (Standard Deviation); unit: years] | 64.6 (12.3) | 65.0 (12.5) | 64.7 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 56 | 93
  Male | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Italy | 38 | 56 | 94

OUTCOME MEASURES:

1. Primary Outcome: Drainage Volume
Description: volume in milliliters of axillary drainage
Time Frame: discharge day
Population: the number of participants for analysis was determined by mean of power sample size calculation
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Ultrasonic | Conventional
Number analyzed (Participants) | 38 | 56
milliliters | 182.6 (267.1) | 525.2 (629.0)
Statistical Analysis 1: Comparison: Ultrasonic vs Conventional; null hypothesis is that drainage volumes are not different; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Time of Discharge
Description: evaluation about the time of discharge from hospital
Time Frame: days
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Ultrasonic | Conventional
Number analyzed (Participants) | 38 | 56
Days | 4.5 (2.1) | 8.1 (5.1)
Statistical Analysis 1: Comparison: Ultrasonic vs Conventional; null hypothesis is that Stay in Hospital Days are not different; Test type: Superiority or Other; p = 0.05, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Ultrasonic | Conventional
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less